CLINICAL TRIAL: NCT05154149
Title: Assessing the Level of Disability and Fear Avoidance Beliefs in Bankers of Karachi
Status: Completed | Type: Observational
Sponsor: Al- Shifa Physiotherapy Institute /Clinic (Other)
Responsible Party: Principal Investigator, Faryal Shoukat, Senior Lecturer, Al- Shifa Physiotherapy Institute /Clinic
Other Study IDs: FShoukat
Record Dates: First submitted 2021-11-26; First posted 2021-12-10 (Actual); Last update posted 2021-12-10 (Actual); Status verified 2021-12

CONDITIONS: Neck Pain
Keywords: Fear Avoidance Belief; musculoskeletal Disorders; neck pain
MeSH Terms: conditions — Neck Pain; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Neck Disability Pain Index — Single time collection of the data

SUMMARY:
An observational study will be conducted to determine the level of pain and disability among bankers working in different banking setups for past 2 years by using Neck Disablity Pain Index and Fear Avoidance Belief Questionnaire. the participant will be recruted fromdifferent private and public banking sectors of Karachi, including Habib bank limited, Silk bank,JS bank and other.

DETAILED DESCRIPTION:
A cross-sectional study with a total sample size of 100 participants will be recruited for the purpose of the survey. The participants will be given Neck Disability Pain Index Questionnaire and Fair avoidance belief Questionnaire in order to determine the level of pain and disability among bankers who are performing their duties in bank from atleast two years.

ELIGIBILITY:
Inclusion Criteria:

* bankers with neck pain

Exclusion Criteria:

* neck surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Bankers with neck pain working in the bank for past two years
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-09-20 (Actual)

PRIMARY OUTCOMES:
Neck Disability Pain Index | 4 weeks
  Quantification of pain and disabilty

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Shifa Institute, Hyderābād, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No